CLINICAL TRIAL: NCT04557683
Title: Perioperative Complications of Deep Extubation in Adults Undergoing Head and Neck Surgery at Massachusetts Eye and Ear Infirmary.
Brief Title: Perioperative Complications of Deep Extubation in Adults
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Jeremy Juang, Anesthesiologist, Massachusetts Eye and Ear Infirmary
Other Study IDs: 1047249
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose a prospective observational cohort study in order to investigate the perioperative respiratory complications of deep extubation in adults undergoing eye and head-and-neck surgery at Massachusetts Eye and Ear. Data pertaining to perioperative respiratory complications from adult patients presenting to MEE for eye and head and neck surgery who undergo deep extubation will be collected for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who present to MEE for eye and head-and-neck surgery and undergo deep extubation will be included.

Exclusion Criteria:

* The study does not exclude anyone from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Based on previous published study by Asai et al, the investigators proposed that a sample size of 300 patients will enable the group to report the complication rates with adequate precision in terms of a sufficiently narrow two-sided 95% confidence interval. Potentially eligible subjects for this study are all adult patients who undergo eye and head-and-neck surgery as well as deep extubation at the end of the surgery per the discretion of the anesthesiologist assigned to the case. Deep extubation is the default extubation method practiced at MEE. Therefore, there will be a sufficient number of potentially eligible subjects to meet the target enrollment goals.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Desaturation | 1 hour
  Desaturation to less than 95% for more than 10 seconds;
Cough | 1 hour
  Episodes of persistent cough, defined as 3 or more consecutive coughs
Laryngospasm | 1 hour
  Episodes of complete or partial laryngospasm
Bronchospasm | 1 hour
  Episodes of bronchospasm
Negative pressure pulmonary edema | 1 hour
  Incidence of negative pressure pulmonary edema
Interventions | 1 hour
  Obstruction that requires intubation or maneuvers, oral airway or jaw thrust

SECONDARY OUTCOMES:
Length of time from the end of surgery to leaving the OR | 1 hour

OTHER OUTCOMES:
Length of stay from admission to the PACU to discharge home | 1-3 hours
Any unplanned hospital admission due to perioperative respiratory adverse events | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Martha Cordoba, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

REFERENCES:
- [Background] Miller KA, Harkin CP, Bailey PL. Postoperative tracheal extubation. Anesth Analg. 1995 Jan;80(1):149-72. doi: 10.1097/00000539-199501000-00025. No abstract available. PMID 7802273
- [Background] Hartley M, Vaughan RS. Problems associated with tracheal extubation. Br J Anaesth. 1993 Oct;71(4):561-8. doi: 10.1093/bja/71.4.561. No abstract available. PMID 8260307
- [Background] Asai T, Koga K, Vaughan RS. Respiratory complications associated with tracheal intubation and extubation. Br J Anaesth. 1998 Jun;80(6):767-75. doi: 10.1093/bja/80.6.767. PMID 9771306
- [Background] von Ungern-Sternberg BS, Davies K, Hegarty M, Erb TO, Habre W. The effect of deep vs. awake extubation on respiratory complications in high-risk children undergoing adenotonsillectomy: a randomised controlled trial. Eur J Anaesthesiol. 2013 Sep;30(9):529-36. doi: 10.1097/EJA.0b013e32835df608. PMID 23344124

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04557683/Prot_SAP_000.pdf